CLINICAL TRIAL: NCT02018718
Title: Development and Validation Phase of Diffusion Tensor Imaging and Arterial Spin Labelling at 3 Tesla Using a Long-term Effort Model Applicable to Skeletal Muscle Characterization.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9097
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2013-12

CONDITIONS: Marathoners
Keywords: Skeletal muscle; Marathon; MRI
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Marathoners (Other)
  Interventions: Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI)

SUMMARY:
The aim of this study is to demonstrate and quantify the micro architecture and micro vascular changes within skeletal muscles after marathon using 3T MRI (diffusion tensor and arterial spin labeling). Apparent diffusion coefficient, fractional anisotropy and flow parameters will be registered before and after the long-distance run on the lower leg. Axial T1 and axial SPAIR sequences will also be applied at the same time.Stress ox and inflammatory markers will be collected in blood and urine samples and compare with both MRI and Near-infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

* Realizing between 2:10 and 4:30 in the marathon.

Exclusion Criteria:

* Smoker
* Subject with medical treatment or with a treatment interrupted for less than 30 days.
* Subject with a osteo-articular, cardiovascular, infectious, lung pathology and/or a metabolic chronic pathology.
* MRI Contraindication : Claustrophobic subject ; subject with a intra-cranial vascular clip, with a pacemaker, with a neurostimulator or a cochlear implant ; subject with intraocular metallic foreign bodies.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Fractional Anisotropy (FA) measure | at 4 days
  The measures will be made from sequences echoplanar (EAR), and will be extracted by post-treatment software Siemens untitled " Syngo" and "FSL", allowing a distortions correction.

SECONDARY OUTCOMES:
Apparent Diffusion Coefficient (ADC) value | at 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien BOMMART, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France